CLINICAL TRIAL: NCT00686634
Title: Sitagliptin in Combination Oral Agent Therapy for Type 2 Diabetes
Brief Title: Sitagliptin in Combination With Metformin and Sulfonylurea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charles Drew University of Medicine and Science (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-06-002; U54RR014616 (NIH)
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Results first posted 2014-11-26 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: sitagliptin; type 2 diabetes; combination therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Sitagliptin 100 mg once daily
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin 100 mg by mouth once daily
  Other Names: Trade name: Januvia

SUMMARY:
This study will compare the effect of a new oral agent for type 2 diabetes, sitagliptin, in comparison to thiazolidinediones as the third-line oral agent, in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
The aim of this protocol is to determine the non-inferiority of the effectiveness of sitagliptin compared to a control group of patients treated with thiazolidinediones as add-on therapy, in low-income ethnic minority type 2 diabetic patients who are failing to maintain adequate control with maximal doses of metformin and a sulfonylurea agent.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18-75
* Type 2 diabetes
* At least 3 months of treatment with maximum tolerated doses of metformin and a sulfonylurea agent, and inadequate glycemic control (Hemoglobin A1c (HbA1c) >7.0%)
* Able to comply with all scheduled visits and requirements of the protocol

Exclusion Criteria:

* Any contraindications to the use of metformin or a sulfonylurea agent
* Extreme hyperglycemia or symptoms of polyuria or polydipsia
* Current or previous chronic use of insulin (other than for treatment of gestational diabetes)
* History of confirmed (or clinical suspicion of) type 1 diabetes mellitus
* Episodes of symptomatic hypoglycemia averaging greater than once per day
* Estimated glomerular filtration rate (eGFR) < 60 mL/min
* Subjects with active hemolytic anemias or hemoglobin variants that render the measurement of HbA1c unreliable
* History of any clinically significant hepatic, cardiovascular (including the use of digoxin), or other major systemic disease that may make the use of sitagliptin unsafe, or otherwise make the interpretation of the data difficult.
* Female subjects of childbearing potential who are sexually active and not using a reliable form of contraception
* Current pregnancy or lactation.
* Subjects who will likely require or initiate therapy with drugs that may interfere with glucose metabolism during the course of the study.
* Subjects who are in another investigational study or have received another investigational medication within 30 days of study entry
* Subjects who are unable or unwilling to give informed consent, comply with all components of the study protocol, attend all scheduled follow-up visits, or present other barriers that would make the implementation of the protocol unusually difficult.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2008-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Hsia, MD, Principal Investigator — Charles Drew University of Medicine and Science
Locations (1):
- Charles Drew University of Medicine and Science, Los Angeles, California, United States

REFERENCES:
- [Derived] Hsia SH, Navar MD, Duran P, Shaheen M, Davidson MB. Sitagliptin compared with thiazolidinediones as a third-line oral antihyperglycemic agent in type 2 diabetes mellitus. Endocr Pract. 2011 Sep-Oct;17(5):691-8. doi: 10.4158/EP10405.OR. PMID 21550951

RESULTS

PARTICIPANT FLOW:
Groups:
- Sitagliptin Treatment: Sitagliptin 100 mg orally once daily
Period: Overall Study
Arm/Group | Sitagliptin Treatment
Started | 108
Completed | 102
Not Completed | 6
Not completed — Protocol Violation | 6

BASELINE CHARACTERISTICS:
Groups:
- Sitagliptin Treatment: Sitagliptin 100 mg once daily
Arm/Group | Sitagliptin Treatment
Number analyzed (Participants) | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 104
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 40
Region of Enrollment [Number; unit: participants]
  United States | 108

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c (HbA1c) Change From Baseline
Time Frame: Baseline, 4 months
Population: Last Observation Carried Forward for subjects with paradoxical worsening of control (switched to alternate treatment before 4 months)
Measure: Mean (Standard Deviation); unit: percentage
Groups:
- Sitagliptin: Sitagliptin 100 mg daily
Arm/Group | Sitagliptin
Number analyzed (Participants) | 102
percentage | -1.3 (1.8)

2. Secondary Outcome: Number of Subjects With Hemoglobin A1c 7.5% or Less at 4 Months
Time Frame: 4 months
Measure: Number; unit: participants
Arm/Group | Sitagliptin
Number analyzed (Participants) | 102
participants | 47

3. Secondary Outcome: Number of Subjects Maintaining Hemoglobin A1c 7.5% or Less by 1 Year
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Sitagliptin
Number analyzed (Participants) | 44
participants | 26

4. Secondary Outcome: Number of Adverse Events
Time Frame: 1 year
Measure: Number; unit: Adverse event
Groups:
- Sitagliptin: Any adverse events while receiving sitagliptin
Arm/Group | Sitagliptin
Number analyzed (Participants) | 108
Adverse event
  Hypoglycemia | 3
  Other adverse events | 3

ADVERSE EVENTS:
Arm/Group | Sitagliptin Treatment
Serious Adverse Events (participants affected / at risk) | 0/108
Other Adverse Events (participants affected / at risk) | 0/108

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes